CLINICAL TRIAL: NCT07069270
Title: A Prospective, Single-center, Single-arm Clinical Study of Adebrelimab in Combination With Vunakizumab and Chemotherapy as First-line Treatment for Extensious-stage Small Cell Lung Cancer
Brief Title: A Study on the First-line Treatment of Small Cell Lung Cancer With Adebrelimab and Vunakizumab and Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2025-218-01
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Vunakizumab; Adebrelimab; Small Cell Lung Cancer
Keywords: Small cell lung cancer; Adebrelimab; Vunakizumab
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab in combination with Vunakizumab and chemotherapy (Experimental)
  Interventions: Drug: Vunakizumab (IL-17A inhibitor); Drug: Adebrelimab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Vunakizumab (IL-17A inhibitor) — Vunakizumab , 240mg, D1, subcutaneous injection, Q4W.
Drug: Adebrelimab — Adebrelimab, 1200 mg, D1, intravenous drip, Q3W
Drug: Chemotherapy — Etoposide, 100mg /m², D1-3, IV, Q3W. Carboplatin, AUC 5, D1, IV, Q3W

SUMMARY:
This study is a prospective, single-center, single-arm clinical trial, with a planned enrollment of 28 cases.The first Adebrelimab +Vunakizumab +EC was administered within 72 hours after enrollment for 4 to 6 cycles.At the end of the combination phase, non-PD subjects entered the maintenance treatment period of Adebrelimab plus Vunakizumab.Treatment will continue until any of the following situations occur: disease progression in the subject, intolerable toxic and side effects, comorbidiments that affect further treatment, the investigator's decision to withdraw the subject from the study, or other reasons for non-compliance with the study treatment or the study procedures or protocols.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 to 75 years old, both male and female are acceptable.
* 2. Histologically or cytologically confirmed extensive-stage small cell Lung cancer (according to the Veterans Administration Lung Study Group, VALG staging);
* 3. No previous systematic treatment;
* 4. Life expectancy exceeds 3 months;
* 5.ECOG physical condition score: 0 to 1 point;
* 6. According to the RECIST 1.1 standard, the target lesion has at least one measurable diameter.
* 7. Within one week before enrollment, the functions of important organs met the following criteria:

  1. blood routine: white blood cell count (WBC) ≥ 3.0 × 109/L; absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelet (PLT) ≥ 100 × 109/L; The hemoglobin content (HGB) is ≥ 9.0 g/Dl
  2. Liver function: aspartate transferase (AST) ≤ 2.5 × ULN, alanine aminotransferase (ALT) ≤ 2.5 × ULN For subjects with liver metastases, their ALT and AST levels were ≤ 5 × ULN. Serum total bilirubin (TBIL) ≤ 1.5 × ULN (except for Gilbert syndrome ≤ 3 × ULN); albumin (ALB) ≥ 30.0 g/L
  3. Renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CrCl) ≥ 50 mL/minute (using the Cockcroft/Gault formula)
  4. Coagulation function: The international normalized ratio (INR) is ≤ 1.5, and the activated partial thromboplastin time (APTT) is ≤ 1.5 × ULN
  5. Others: Lipase ≤ 1.5 × ULN. If the lipase is greater than 1.5 × ULN and there is no clinical or radiological confirmation of pancreatitis, the patient can be enrolled. Amylase ≤ 1.5 × ULN. If the amylase is greater than 1.5 × ULN and there is no clinical or radiological confirmation of pancreatitis, the patient can be enrolled. alkaline phosphatase (ALP) ≤ 2.5 × ULN, for bone metastasis subjects, ALP ≤ 5 × ULN
  6. Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥ 50%;
* 8.Women of childbearing age must undergo a serum pregnancy study within 7 days before the first medication, and the result must be negative. Female subjects of childbearing age and male subjects whose partners are women of childbearing age must agree to contraception from the signing of the informed consent form until 24 weeks after the last administration of the study drug.
* 9. The subjects voluntarily joined this study, signed the informed consent form, had good compliance and cooperated with the follow-up.

Exclusion Criteria:

* 1. There is a large amount of uncontrolled pleural effusion, pericardial effusion or ascites;
* 2. The following heart disorders exist: (1) According to NYHA cardiac function classification, (1) Grade III-IV cardiac function; (2) Unstable angina pectoris or acute ischemia indicated by electrocardiogram or myocardial infarction occurred within one year; (3) Clinically significant supraventricular or ventricular arrhythmias and other conduction system abnormalities (including QTc interval ≥ 450ms in men and ≥470ms in women); (4) Clinically significant pericardial and myocardial diseases.
* 3. Insufficient bone marrow reserve or organ function;
* 4. Systemic immunomodulators (including but not limited to thymosin, interferon or interleukin-2) have been used for treatment within 4 weeks before enrollment;
* 5. Corticosteroid hormones (> 10 mg/ day prednisone or equivalent dose) or other immunosuppressants were used within 2 weeks before enrollment;
* 6. Have any active autoimmune diseases or a history of autoimmune diseases; Interstitial pneumonia, drug-induced pneumonia, radiation pneumonitis requiring steroid treatment, or active pneumonia with clinical symptoms;
* 7. There was an active or uncontrolled severe infection (CTCAE 5.0 ≥ grade 2) within 2 weeks before enrollment, and/or received antibiotic treatment;
* 8. Tuberculosis patients who are active or undergoing treatment;
* 9. Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg), history of hypertensive crisis or hypertensive encephalopathy;
* 10. Within 24 weeks before enrollment, there were hyperactive/venous thrombotic events, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
* 11. Has undergone invasive surgery within 4 weeks before enrollment;
* 12. Positive for HBsAg and HBV DNA test value exceeding the upper limit of the normal reference value (1000 copies /mL or 100 IU/mL), or positive for HCV (HCV RNA or HCV Ab test indicating acute or chronic infection), or a history of HIV positivity;
* 13. Patients who have received live vaccines within 12 weeks before enrollment;
* 14. Known to be allergic to the research drug or excipients, and known to have a severe allergic reaction to any monoclonal antibody;
* 15. A known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* 16. Other malignant tumors concurrent within 5 years before enrollment are excluded, except for fully treatable cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and ductal carcinoma in situ after radical resection.
* 17. It is known that there are serious mental disorders, alcoholism, drug abuse or drug abuse, etc.
* 18. Have received any other investigational drug treatment or participated in another interventional clinical study within 4 weeks prior to signing the ICF;
* 19. As determined by the researchers, the subjects have other factors that may lead to the forced termination of this study, such as non-compliance with the protocol, other serious diseases (including mental disorders) requiring concurrent treatment, severe laboratory test abnormalities, accompanied by family or social factors that may affect the safety of the subjects, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
12-month PFS rate | 12-month

SECONDARY OUTCOMES:
Progression-free survival (PFS） | 12- months
Overall survival (OS） | 24-months
Objective response rate (ORR） | Each 2 cycles can last up to 3 months (each cycle is 21 days).
Disease Control Rate (DCR） | Each 2 cycles can last up to 3 months (each cycle is 21 days).
The incidence and severity of adverse events (AE) and serious adverse events (SAE) | As long as two years